CLINICAL TRIAL: NCT01510938
Title: Role of Probiotics in Prevention of Respiratory Tract Infections in Preschool and Primary School Children
Brief Title: Probiotics in Respiratory Tract Infections in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Sergei V. Gerasimov, MD, PhD, Associate Professor of Pediatrics, Lviv National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SG-11009
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Infections, Respiratory Tract
Keywords: Children; Respiratory Tract Infections; Prevention
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1 g of rice maltodextrin will be reconstituted in 25-50 ml of tepid water or juice and immediately fed once a day for 2-weeks trial period or to the end of acute respiratory infection depending on whatever is longer.
  Interventions: Dietary Supplement: Placebo
- Probiotic (Experimental): powder of L. acidophilus DDS-1, B. lactis UABLA-12, 50 mg of fructooligosaccharide
  1 g of probiotic will be reconstituted in 25-50 ml tepid water or juice and immediately fed once a day (5 billion CFU/daily) for 2-weeks trial period or to the end of acute respiratory infection depending on whatever is longer.
  Interventions: Dietary Supplement: L. acidophilus DDS-1, B. lactis UABLA-12

INTERVENTIONS:
Dietary Supplement: L. acidophilus DDS-1, B. lactis UABLA-12 — 1 g of probiotic will be reconstituted in 25-50 ml tepid water, juice or age specific baby food and immediately fed once a day (5 billion CFU/daily) for 2-weeks trial period or to the end of acute respiratory infection depending on whatever is longer.
  Other Names: DDS-Junior
  Arms: Probiotic
Dietary Supplement: Placebo — 1 g in 25-50 ml of tepid water or juice fed once a day for 2-weeks trial period or to the end of acute respiratory infection depending on whatever is longer.
  Other Names: Rice maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the potential of probiotics in prevention of respiratory tract infections and their complications in children

ELIGIBILITY:
Inclusion Criteria:

* Age 3-12 yrs
* At least one episode of respiratory tract infection in the previous epidemiological season
* Direct telephone access available
* Informed consent signed

Exclusion Criteria:

* Vaccination against the influenza
* Chronic adeno-tonsillar pathology
* Recurrent otitis
* Sinusitis
* Respiratory allergy
* Acute or chronic intestinal disease with diarrhea and/or malabsorption syndrome
* Lactose intolerance
* Functional or organic constipation
* Down syndrome
* Congenital or acquired heart disease
* Cerebral palsy
* Any chronic hepatic, renal, metabolic, or immune system disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory tract infection episodes in a child | 1 month
  An episode will be defined as display of fever, cough, rhinitis, and sore throat or combination thereof for longer than 48 hours

SECONDARY OUTCOMES:
Duration of respiratory tract infection | 21 days
  Time to CARIFS (Canadian Acute Respiratory Illness and Flu Scale) value 0
Severity of respiratory tract infection | 21 days
  a product of daily CARIFS times the duration of the disease
Complications of respiratory tract infections | 21 days
  Percent of otitis, sinusitis, bronchitis, pneumonia cases
Antibiotic prescriptions | 21 days
  Percent
Hospitalization rate | 21 days
  Number of hospitalizations
Number of unscheduled doctor visits | 21 days
Number of days daycare/school missed | 21 days
Number of workdays missed by parents | 21 days
Time to resolution of individual CARIFS item | 21
  Days to the correspondent CARIFS item 0
25% and 50% decrease in the CARIFS score | 21day
  25% and 50% decrease in the CARIFS score
Percent and duration of the use of over-the-counter medications | 21day
  Percent and duration of the use of over-the-counter medications

CONTACTS AND LOCATIONS:
Overall Officials: Sergei V Gerasimov, M.D., Ph.D., Principal Investigator — Lviv National Medical University
Locations (1):
- Lviv City Children Hospital, Lviv, Lviv Oblast, Ukraine